CLINICAL TRIAL: NCT04011371
Title: Cyanoacrylate Closure for Treatment of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 424-2017
Record Dates: First submitted 2019-07-05; First posted 2019-07-08 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyanoacrylate closure (Experimental): Subjects enrolled in the study will undergo ultrasound guided vein closure using the VenaSealTM cyanoacrylate delivery device.
  Interventions: Procedure: Cyanoacrylate closure

INTERVENTIONS:
Procedure: Cyanoacrylate closure — Cyanoacrylate glue embolization targeting venous insufficiency

SUMMARY:
Venous leg ulcers (VLUs) are a common wound with significant morbidity and cost, and suboptimal therapeutic options. VLUs result from chronic venous insufficiency, including venous reflux and post-thrombotic syndrome. VLU can take from months to years to heal, and 54-78% recur. Current therapies include wound, compression therapy, and medications. These treatments can increase the rate of healing, and reduce recurrence, however these therapies can be burdensome, painful, and ineffective, and despite these therapies, ~50% of wounds become chronic. Chronic VLUs can be painful, malodorous, and infected, and they often significantly limit an individual's function and mobility. An emerging therapy for symptomatic venous reflux is the closure of the culprit vein by endovenous closure with a cyanoacrylate adhesive implant. Recent studies show cyanoacrylate closure (CAC) to be a safe and effective treatment for varicosities resulting from symptomatic incompetent great saphenous veins. This study will evaluate the safety and effectiveness of CAC for VLUs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old at time of screening;
2. Venous leg ulcer;
3. Venous insufficiency (>0.5 seconds; confirmed by Doppler within last 6 months);
4. ABI of ≥0.9;
5. Capable of understanding the study and providing informed consent.

Exclusion Criteria:

1. Previous hypersensitivity reactions to the VenaSealTM adhesive or cyanoacrylates;
2. Acute superficial thrombophlebitis;
3. Bilateral treatment
4. Thrombophlebitis migrans;
5. Deep venous thrombosis;
6. Deep venous incompetence or occlusion in external iliac or distal veins in the affected extremity (as assessed based on spontaneity, phasicity, augmentation, pulsatility, and compressibility on ultrasound);
7. Post-thrombotic syndrome;
8. Acute sepsis;
9. Coagulation disorders;
10. Radiation or chemotherapy within 3 months of study;
11. Pregnant or lactating females;
12. Uncontrolled diabetes (HbA1c >10%);
13. Diabetic foot ulcers;
14. Current use of systemic anticoagulation;
15. Previous treatment of target vein;
16. Tortuous veins;
17. Current participation in another interventional study, or participation within 30 days prior to screening;
18. Inability to tolerate compression, or to receive endovenous treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events | 3 months
Healing rate | 3 months
  Change in ulcer size

SECONDARY OUTCOMES:
Rate of adverse events | 12 months
Healing rate | 12 months
  Change in ulcer size
Closure rate | 12 months
  Time to ulcer closure
Patient-reported quality of life: EuroQol Five Dimension Scale: EQ-5D-5L Health Questionnaire | 12 months
  EuroQol Five Dimension Scale: EQ-5D-5L Health Questionnaire - measures patient-reported health related to five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses for each parameter are coded 1-5, with a lower score reflecting better health, and a higher score meaning worse health. Overall health is self-rated on a scale 0-100, with 0 meaning the worst and 100 meaning the best health imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Callam MJ. Epidemiology of varicose veins. Br J Surg. 1994 Feb;81(2):167-73. doi: 10.1002/bjs.1800810204. PMID 8156326
- [Result] Fowkes FG, Evans CJ, Lee AJ. Prevalence and risk factors of chronic venous insufficiency. Angiology. 2001 Aug;52 Suppl 1:S5-15. doi: 10.1177/0003319701052001S02. PMID 11510598
- [Result] Van den Oever R, Hepp B, Debbaut B, Simon I. Socio-economic impact of chronic venous insufficiency. An underestimated public health problem. Int Angiol. 1998 Sep;17(3):161-7. PMID 9821029
- [Result] Abbade LP, Lastoria S. Venous ulcer: epidemiology, physiopathology, diagnosis and treatment. Int J Dermatol. 2005 Jun;44(6):449-56. doi: 10.1111/j.1365-4632.2004.02456.x. PMID 15941430
- [Result] Olin JW, Beusterien KM, Childs MB, Seavey C, McHugh L, Griffiths RI. Medical costs of treating venous stasis ulcers: evidence from a retrospective cohort study. Vasc Med. 1999;4(1):1-7. doi: 10.1177/1358836X9900400101. PMID 10355863
- [Result] Mayer W, Jochmann W, Partsch H. [Varicose ulcer: healing in conservative therapy. A prospective study]. Wien Med Wochenschr. 1994;144(10-11):250-2. German. PMID 7856198
- [Result] Bergqvist D, Lindholm C, Nelzen O. Chronic leg ulcers: the impact of venous disease. J Vasc Surg. 1999 Apr;29(4):752-5. doi: 10.1016/s0741-5214(99)70330-7. No abstract available. PMID 10194512
- [Result] Evans CJ, Fowkes FG, Ruckley CV, Lee AJ. Prevalence of varicose veins and chronic venous insufficiency in men and women in the general population: Edinburgh Vein Study. J Epidemiol Community Health. 1999 Mar;53(3):149-53. doi: 10.1136/jech.53.3.149. PMID 10396491
- [Result] Lazarus GS, Cooper DM, Knighton DR, Percoraro RE, Rodeheaver G, Robson MC. Definitions and guidelines for assessment of wounds and evaluation of healing. Wound Repair Regen. 1994 Jul;2(3):165-70. doi: 10.1046/j.1524-475X.1994.20305.x. PMID 17156107
- [Result] Kelechi TJ, Johnson JJ, Yates S. Chronic venous disease and venous leg ulcers: An evidence-based update. J Vasc Nurs. 2015 Jun;33(2):36-46. doi: 10.1016/j.jvn.2015.01.003. PMID 26025146
- [Result] Morrison N, Gibson K, McEnroe S, Goldman M, King T, Weiss R, Cher D, Jones A. Randomized trial comparing cyanoacrylate embolization and radiofrequency ablation for incompetent great saphenous veins (VeClose). J Vasc Surg. 2015 Apr;61(4):985-94. doi: 10.1016/j.jvs.2014.11.071. Epub 2015 Jan 31. PMID 25650040
- [Result] Almeida JI, Javier JJ, Mackay E, Bautista C, Proebstle TM. First human use of cyanoacrylate adhesive for treatment of saphenous vein incompetence. J Vasc Surg Venous Lymphat Disord. 2013 Apr;1(2):174-80. doi: 10.1016/j.jvsv.2012.09.010. Epub 2012 Dec 22. PMID 26992340
- [Result] Proebstle TM, Alm J, Dimitri S, Rasmussen L, Whiteley M, Lawson J, Davies A. Twelve-Month Follow-up of the European Multicenter Study on Cyanoacrylate Embolization of Incompetent Great Saphenous Veins. J Vasc Surg Venous Lymphat Disord. 2014 Jan;2(1):105-6. doi: 10.1016/j.jvsv.2013.10.009. Epub 2013 Dec 12. No abstract available. PMID 26992985